CLINICAL TRIAL: NCT01689545
Title: Prevention for Positives: A Randomized Controlled Trial Among Vietnamese HIV-positive Injecting Drug Users
Brief Title: Prevention for Positives: An RCT Among Vietnamese HIV-positive IDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 5R01DA022962 (NIH)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: HIV
Keywords: HIV; drug abuse; social stigma; Vietnam
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Individual level (Experimental)
  Interventions: Behavioral: Individual level; Behavioral: Structural level standard of care
- Structural level (Experimental)
  Interventions: Behavioral: Structural level; Behavioral: Individual level standard of care
- Combined individual & structural level (Experimental)
  Interventions: Behavioral: Individual level; Behavioral: Structural level
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Individual level standard of care; Behavioral: Structural level standard of care

INTERVENTIONS:
Behavioral: Individual level — Index participants will participate in standard HIV VCT supplemented with 2 posttest counseling sessions, followed by 2 post-test skill-building support groups for HIV positive IDUs.
  Arms: Combined individual & structural level; Individual level
Behavioral: Structural level — Community members will participate in 2 community-based HIV and IDU stigma videos combined with a series of visits with community outreach workers.
  Arms: Combined individual & structural level; Structural level
Behavioral: Individual level standard of care — The education materials that are currently offered in Thai Nguyen will be delivered didactically by health workers on 1) the HIV situation in Vietnam; 2) consequences of drug use; 3) routes of HIV transmission; and 4) options for drug treatment.
  Arms: Standard of Care; Structural level
Behavioral: Structural level standard of care — Posters and billboards on HIV/AIDS transmission, leaflets on HIV/AIDS transmission available in health station, 15-minute monthly public broadcasts (via the village loudspeaker) on the consequences of HIV/AIDS and the number of HIV cases in the country and province will be delivered in communities.
  Arms: Individual level; Standard of Care

SUMMARY:
The purpose of this study is to determine whether a combined individual and structural level stigma reduction intervention is effective in reducing high risk injecting and sexual behaviors among HIV positive injecting drug users.

DETAILED DESCRIPTION:
This study is a randomized controlled trial among HIV-positive injecting drug users (IDUs) to reduce high risk injecting and sexual behaviors in Thai Nguyen, Vietnam. We will be conducting this study in collaboration with the Thai Nguyen Centre for Preventive Medicine (CPM). We will compare standard HIV voluntary counseling and testing (VCT) to an intervention that adds a continuum of psychosocial support for HIV-positive IDUs. The intervention consists of a two-tiered approach that addresses structural and individual level barriers to risk reduction: 1) The structural level of the intervention consists of community-based programs and targets HIV stigma that is a primary obstacle to risk reduction for HIV-positive individuals; 2) The individual level of the intervention consists of 2 HIV posttest counseling sessions and 2 skill-building support groups for HIV-positive IDUs. Our research questions for the overall project are:

1. What is the impact of perceived HIV-related stigma on disclosure, social support, and coping among IDUs?
2. What roles do disclosure, social support, and coping play in facilitating the reduction of HIV-risk behaviors
3. Are combined individual and structural level interventions more effective in reducing injecting and sexual behaviors among HIV-positive IDUs than individual or structural interventions alone and more effective than the standard HIV VCT?

ELIGIBILITY:
Index participant

Inclusion Criteria:

* laboratory confirmed HIV positive diagnosis
* able and wiling to bring an injecting network member for screening
* injected drugs in previous 6 months
* planned residence in Thai Nguyen for next 24 months

Exclusion Criteria:

* unwilling to provide locator information
* unable to participate in group counseling sessions due to psychological disturbance, cognitive impairment or threatening behavior
* currently participating in other HIV or drug use intervention activities

Network member participant

Inclusion Criteria:

* laboratory confirmed HIV negative diagnosis
* injected or shared drug paraphernalia in past 6 months
* interacts at least once a week with index participant

Exclusion Criteria:

* unwilling to provide locator information
* having psychological or cognitive impairment
* currently participating in other HIV intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2175 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
HIV injecting risk behavior | 2 years
  Change in self-reported use of new injecting equipment
HIV sexual risk behavior | 2 years
  Change in self-reported condom use during sexual intercourse

SECONDARY OUTCOMES:
HIV incidence | 2 years
  Change in HIV incidence among network members

OTHER OUTCOMES:
Perceived HIV-related stigma | 2 years
  Change in self-reported perceived HIV-related stigma among index participants

CONTACTS AND LOCATIONS:
Overall Officials: Vivian F Go, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Preventive Medicine, Thái Nguyên, Thai Nguyen, Vietnam

REFERENCES:
- [Derived] Levintow SN, Pence BW, Powers KA, Sripaipan T, Ha TV, Chu VA, Quan VM, Latkin CA, Go VF. Estimating the Effect of Depression on HIV Transmission Risk Behaviors Among People Who Inject Drugs in Vietnam: A Causal Approach. AIDS Behav. 2021 Feb;25(2):438-446. doi: 10.1007/s10461-020-03007-9. PMID 32833193
- [Derived] Levintow SN, Pence BW, Ha TV, Le Minh N, Sripaipan T, Latkin CA, Vu PT, Quan VM, Frangakis C, Go VF. Depressive Symptoms at HIV Testing and Two-Year All-Cause Mortality Among Men Who Inject Drugs in Vietnam. AIDS Behav. 2019 Mar;23(3):609-616. doi: 10.1007/s10461-018-2318-8. PMID 30357641
- [Derived] Go VF, Frangakis C, Minh NL, Latkin C, Ha TV, Mo TT, Sripaipan T, Davis WW, Zelaya C, Vu PT, Celentano DD, Quan VM. Efficacy of a Multi-level Intervention to Reduce Injecting and Sexual Risk Behaviors among HIV-Infected People Who Inject Drugs in Vietnam: A Four-Arm Randomized Controlled Trial. PLoS One. 2015 May 26;10(5):e0125909. doi: 10.1371/journal.pone.0125909. eCollection 2015. PMID 26011427